CLINICAL TRIAL: NCT04893135
Title: Impact of the Rapid Normalization of Chronic Hyperglycemia and the Practice of Moderate Physical Activity on the "Receptor Activator of Nuclear Factor-kappa B Ligand / Osteoprotégérine (RANKL / OPG) System in Patients Living With Type II Diabetes
Acronym: RANKL-GLYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRCB 2021-A00576-35
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Type II Diabetes
Keywords: Diabetes's complications; neuroarthropathy Physical activity; RNKL/OPG
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1A (No Intervention): Uncontrolled diabetes (HbA1c> 8.5%) over 6 months. In order to assess the effect of rapid correction of HbA1c on RANKL levels, without the practice physical activity
- G1B (Experimental): Uncontrolled diabetes (HbA1c> 8.5%) over 6 months. In order to assess the effect of rapid correction of HbA1c on RANKL levels, with the practice physical activity
  Interventions: Other: pratice physical activity
- G2 (No Intervention): Controlled diabetes (HbA1c level <7%). This group will study the natural course of RANKL levels in balanced diabetic patients.

INTERVENTIONS:
Other: pratice physical activity — treadmill walking : walk at a speed of 2.7 km.h-1 in 3 stages of 3 mins with an incline of 0%, 5% and 10%
  Arms: G1B

SUMMARY:
The rapid normalization of hyperglycemia can cause a neuropathy called Diabetes Treatment-Induced Neuropathy (NITD). This phenomenon induces the presence of hyper vascularization and inflammation in contact with the nerve ends.

In another register in patients living with diabetes, it has been observed the development of a rare and devastating complication for the joints called the so-called neuroarthropathy of Charcot (CN).

DETAILED DESCRIPTION:
The rapid normalization of hyperglycemia can cause a neuropathy called Diabetes Treatment-Induced Neuropathy (NITD). This phenomenon induces the presence of hyper vascularization and inflammation in contact with the nerve ends.

In another register in patients living with diabetes, it has been observed the development of a rare and devastating complication for the joints called the so-called neuroarthropathy of Charcot (CN). The pathophysiology of CN is not completely known but there is an activation of markers of inflammation and bone remodeling, disruption of the osteoblast and osteoclast system, activation of the RANKL system (Receptor activator of nuclear factor-kappa B ligand) and its antagonist osteoprogesterin (OPG). Inflammation and peripheral hypervascularization therefore seem to be a common link between the two pathologies mentioned (NITD and CN). We have confirmation that the rapid correction of chronic hyperglycemia can trigger (not systematically) NITD, but what about the influence of this rapid correction on the appearance of CN. Furthermore, physical activity (PA) and exercise have long been recognized as the cornerstones of the prevention and management of chronic diseases, due to their beneficial effects on the clinical parameters of various diseases. The practice of PA has a preventive and therapeutic effect against osteoporosis (a disease in which the level of RANKL is particularly high), so there is in theory a preventive effect of the practice of physical activity on the development of CN.

ELIGIBILITY:
Inclusion Criteria:

Group G1:

* Male or female patient aged 18 to 70, not practicing regular physical activity (Baecke score <10)
* Patient with type 2 diabetes for at least 1 year
* Patient treated with metformin +/- SU +/- DPP4 inhibitor +/- GLP1 analogue +/- insulin therapy
* Patient insufficiently balanced under his current treatment with an HbA1c level> 8.5% for 6 months.
* Patient able to practice physical activity on a regular basis
* Patient having performed a coronary artery disease screening test in the year prior to inclusion
* Woman of childbearing age with effective contraception put in place and monitored throughout the trial
* Patient having given his consent to participate in the study and having signed an informed consent
* Within the G1 group, a controlled 1: 1 randomization, stratified on age (≤65 years or> 65 years) and BMI (≤ 30 or> 30) will determine the inclusion of patients in the G1A group (correction of HbA1c) or G1B (correction of HbA1c + physical activity).

Group G2:

* Male or female patient aged 18 to 70, not practicing regular physical activity
* Patient with type 2 diabetes for at least 1 year
* Patient treated with metformin +/- SU +/- DPP4 inhibitor +/- GLP1 analogue +/- insulin therapy
* Patient balanced under his current treatment with an HbA1c level <7% for 6 months.
* Women of childbearing potential with effective contraception put in place and monitored throughout the trial
* Patient having given his consent to participate in the study and having signed an informed consent
* Matching with the last patient included in group G1 on age (± 5 years), sex, duration of diabetes (± 2 years) and BMI (± 2kg / m2).

Exclusion Criteria:

* Fetal and maternal pathologies requiring maturation Patient with type 1 diabetes
* Patient with regular physical activity
* History of severe cardiovascular pathologies (myocardial infarction, or acute coronary syndrome, or stroke in the past year)
* Patient with a history of severe hypoglycemia in the 6 months preceding entry into the study and / or not experiencing hypoglycemia at all
* Patient pregnant or likely to be
* Severe obesity (BMI> 35kg / m2)
* Other pathologies likely to interfere with the glycemic variation: in particular the use of corticosteroids during the study
* Patient already having Charcot's neuroarthropathy or symptomatic autonomic neuropathy: orthostatic hypotension and / or gastro-paresis
* Patient with preproliferative diabetic retinopathy
* Patient having anti RANKL treatment
* Subject under tutorship or curatorship
* Subject not affiliated to social security.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
RANKL/OPG level | at 3 months
  RANKL/OPG level

SECONDARY OUTCOMES:
Sudoscan measurement | at 3 months
  The Sudoscan non-invasively measures the ability of sweat glands to release chloride ions in response to an electrochemical stimulus on the palms of the hands and soles of the feet, areas with the highest density of sweat glands using four independent electrodes placed on the palms of the hands, soles of the feet which have a high density of sweat glands,

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No